CLINICAL TRIAL: NCT00194740
Title: Taxotere Plus Weekly Navelbine and G-CSF: A Phase II Study in Stage IV Breast Cancer
Brief Title: Taxotere Plus Weekly Navelbine and G-CSF: A Study in Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Julie Gralow, M.D., University of Washington
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 97-5372-A
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-12

CONDITIONS: Breast Neoplasm
Keywords: Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Vinorelbine; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Docetaxel; Drug: Vinorelbine; Drug: Filgrastim

INTERVENTIONS:
Drug: Docetaxel — 60 mg/m2, IV, day 1 of each 21 day cycle
  Other Names: Taxotere
Drug: Vinorelbine — 27.5 mg/m2, IV, days 8 & 15 of each 21 day cycle
  Other Names: Navelbine
Drug: Filgrastim — 5 µg/kg/day s.c., to be administered days 2-21 of each cycle.
  Other Names: G-CSF, Neupogen

SUMMARY:
The two drugs used to treat metastatic breast cancer in this study may perform better when used together than when used separately. The use of another drug that prevents the most common side effect of the two-drug combination permits the delivery of both agents at closer to the "full" dose for either when used alone. We hypothesize that the two-drug combination used with G-CSF support will be more effective and less toxic than other standard regimens for the treatment of metastatic breast cancer.

DETAILED DESCRIPTION:
Preclinical data suggest that there may be synergy between vinorelbine and paclitaxel when the two drugs are used in combination such that the effect of the two together may be better than either alone. Clinical data suggest that the use of concurrent G-CSF with paclitaxel and vinorelbine permits the delivery of both agents at approximately 70% of the "full" dose for either, used alone without G-CSF support, with myelosuppression as the usual dose-limiting toxicity and no unusual or unexpected complications. Encouragingly, 8/20 (40%) patients had objective responses, with three complete remissions (15%) in this program of third-line therapy. Therefore, we now propose to combine docetaxel at about 70% of "full" dose with vinorelbine at 27.5 mg/m2, the "phase II" dose defined in the previous trial. Docetaxel will be given on day 1 followed by vinorelbine on days 8 and 15, with G-CSF to be administered on all days except that of docetaxel administration. The cycle is to be repeated every three weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have stage IV, microscopically-confirmed carcinoma of the breast with histologic slides and/or blocks available for review.
* Patients must have relapse or progression while receiving, or within 12 months of having received, anthracycline-containing (doxorubicin or mitoxantrone) regimen as either adjuvant treatment or therapy for advanced breast cancer. Prior Taxol by 3- or 24-hour infusion is permitted. Patients who have received a maximum dose of anthracycline (greater than 450 mg/m2) are also eligible.
* Patients must have measurable (bidimensionally) or evaluable disease.
* Patients must be 18 or more years of age.
* Patients must have a Karnofsky Performance Status greater than or equal to 70% at screen and on the first day of treatment.
* Patients must have a life expectancy of more than 16 weeks.
* Prior irradiation is permitted, provided that prior irradiation does not exceed 25% of the estimated bone marrow volume and provided that measurable/evaluable disease exists outside the radiation field OR there must be histologic proof of progressive disease within a radiation field.
* Informed consent must be obtained prior to registration.
* Patients must be more than 2 weeks from prior surgery; more than 3 weeks from radiation therapy to the pelvis, spine or long bones; more than 3 weeks from prior chemotherapy (more than 6 weeks for mitomycin C or nitrosureas), or more than 2 weeks from prior hormonal therapy.
* All patients must have appropriate central venous access.

Exclusion Criteria:

Patients are excludes if their:

* Granulocyte count is less than 1,500/mm3.
* Platelet count is less than 100,000/mm3.
* Hemoglobin is less than 9 gm/dl.
* Creatinine is greater than 2.0 mg/dl.
* Total bilirubin is greater than ULN (institutional upper limit of normal)..
* SGOT (AST) and/or SGPT (ALT) is greater than 1.5 x ULN concomitant with alkaline phosphatase greater than 2.5 x ULN.

Patients are excluded if they are:

* In visceral crisis characterized by rapidly progressive hepatic or lymphangitic lung metastases.
* Medically unstable.
* Pregnant or lactating.

Patients are excluded if they have:

* Uncontrolled CNS disease.
* Pre-existing clinically significant peripheral neuropathy except for abnormalities due to cancer.
* Psychological, familial, sociological or geographical conditions which do not permit weekly medical follow-up and compliance with the study protocol.
* Prior therapy with Navelbine.
* Sensitivity to E. Coli-derived proteins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 1997-11; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Response to treatment | Until disease progression
Toxicity of treatment | Until completion of treatment

SECONDARY OUTCOMES:
Time to progression | Until disease progression occurs
Over all survival | Until study is closed

CONTACTS AND LOCATIONS:
Overall Officials: Julie R. Gralow, M.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington/Seattle Cancer Care Alliance, Seattle, Washington, United States